CLINICAL TRIAL: NCT02318017
Title: An Electroencephalography Study of the Effects of Psychostimulants on Dynamic Patterns of Cognitive Task-based Functional Connectivity in Youths With Attention Deficit Hyperactivity Disorder
Brief Title: Psychostimulants Effects on Brain Functional Connectivity in Youth With Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SHEBA-14-1351-IH-CTIL
Record Dates: First submitted 2014-11-18; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Adhd
Keywords: adhd; global network; eeg
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate (Active Comparator): Methylphenidate 0.5mg/kg - once
  Interventions: Drug: Methylphenidate
- Placebo (Placebo Comparator): Placebo - once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Before neurocognitive testing, Methylphenidate/Placebo will be given
  Other Names: MPH
  Arms: Methylphenidate
Drug: Placebo
  Arms: Placebo

SUMMARY:
In the current study, we will administer three widely administered cognitive tasks while simultaneously measuring electroencephalography (EEG) in ADHD patients before and after methylphenidate immediate release (IR) treatment compared to placebo. In addition we will compare the effective connectivity dynamics to normal subjects. Using this novel network analysis approach, we will attempt to address the currently limited cognitive network literature. We will attempt to map the connectivity between the discrete brain regions during the execution of the tasks before and after treatment with methylphenidate IR. Comparison with healthy control subjects will enable us to determine whether the direction of methylphenidate induced changes in brain functioning (in youths with ADHD) will be toward or away from normal connectivity patterns. We will also examine whether network patterns differ between the healthy controls and the ADHD patients.

DETAILED DESCRIPTION:
Research objective:

To examine dynamic patterns of task-evoked network connectivity in ADHD patients before and after methylphenidate IR treatment compared with healthy controls.

Aims:

1. To explore whether patterns of network connectivity differs before and after methylphenidate treatment.
2. To explore whether patterns of network connectivity differs between ADHD patients and healthy subjects.

Methods

Subjects Total number of subjects: 55 age 6-18, the widest age range for representation of pediatric population not including preschoolers. The cross-over study design of this study is best suited for a wide study population age range. Preschoolers will not be included because of incompatibility of the computerized neurocognitive tasks.

35 children and adolescent patients undergoing diagnosis and treatment management for ADHD using computerized cognitive tasks (e.g. CPT) with and without methylphenidate treatment.

20 healthy children and adolescents will be recruited.

Recruitment procedure in the study will be as follows:

1. Parents of patients diagnosed with ADHD will be approached at the attention clinic of the Sheba Medical Center to check whether they wish to participate in the study. It should be emphasized that treatment and follow-up at the clinic will not be affected by the participation or non-participation in the study.
2. E-mail and/or phone contact will be made to parents of patients diagnosed with ADHD from the attention clinic of the Sheba Medical Center. Only parents who confirmed in advance (and regardless of the current study) to contact them by e-mail and / or phone will be contacted.
3. During lectures to the general public, performed by the researchers on the subject of ADHD, the research will be presented and offered for parents of ADHD diagnosed child to participate in the study. Information letter will be sent (study group recruitment add attached) to all who express interest of his son / daughter participation in the study.
4. Recruitment of participants in the control group - recruitment announcement of healthy volunteers will be sent using electronic media and shall be accompanied by an information letter (control group recruitment add- attached).

Study group

Children and adolescents which are being considered for methylphenidate treatment and therefore referred to computerized cognitive tasks with and without methylphenidate IR use as part of their management. The recruitment will be from patients referred to the attention clinic at Edmond and Lilly Safra children's Hospital and diagnosed with ADHD. Patients treated with methylphenidate or under consideration for treatment with methylphenidate will be offered to join the study and will be included in the study after the proper consent forms will be signed by them and their parents. Clinical assessment including semi constructed interview by a psychiatrist as part of the regular management will be made.

Control group Healthy children and adolescents will be recruited after signing the proper consent forms by them and their parents. Public publication of the study will take place for the recruitment of the control group. (e.g posters stating the main study objectives, procedures and the subjects needed characteristics)

Recruitment and payment Subjects' parents will be paid only for carfare and loss of time.

Medication: Subjects from the control group already using methylphenidate will have at least 2 days medication wash out prior to the evaluation day.

Methylphenidate IR will be given as a single dose of 0.5 mg/kg.

Experimental design 1. Demographic measures: General demographics questionnaire - i.e. name, gender, age, country of origin, level of education.

2. Neuropsychiatric and side effects assessment:

1. The DuPaul-Berkley ADHD Rating scale - Hebrew version, will be used at baseline session. (Dupaul GJ 1991)
2. Hebrew version of the schedule for Affective disorders and Schizophrenia for school-aged Children, present and lifetime (K-SADS-PL) (Kaufman et al. 1997).
3. Berkley side effects rating scale (modified Hebrew version) will be administered to parents after methylphenidate-IR/placebo. (Berkley RA 1988)
4. The Strengths and Difficulties Questionnaires (SDQ) - Hebrew version, will be used at baseline session for the control group. (Goodman R 1997)
5. Clinical Global Impression - Severity scale (CGI-S) (Guy W, 1976)
6. Clinical examination including psychiatric interview and assessment for soft neurological signs.

3. EEG testing procedure: A 64 channel ActiveTwo Biosemi EEG system (Biosemi Instrumentations, Amsterdam, Netherlands) will be used to record task-related evoked potentials over the entire scalp. Sampling rate at 1024 Hz. ActiveTwo Biosemi EEG system allows calibration changes which are not required for clinical treatment and is used for research purposes only. The ActiveTwo Biosemi EEG system is not used for outpatient or inpatient clinical use in Israel. In this study we will use the ActiveTwo Biosemi EEG system from the Weizmann institute at Sheba medical center. Subjects will be seated comfortably in a chair and the Biosemi cap put on their head. The 64-scalp electrodes are positioned according to the international 10-20 system. To place the cap, we will measure the distance between the nasion and inion and the distance between the two ears and situated the cap so that electrode Cz was exactly half way between the two ears and between nasion (intersection of the frontal bone and two nasal bones) and inion (external occipital protuberance).

Baseline EEG measure: Prior to the cognitive testing, a baseline EEG recording of 5 minutes will be required to generate a baseline network map of brain connectivity.

Cognitive EEG measure: Throughout the cognitive testing (detailed below), EEG will be recording the neural response and the data will be processed offline.

4. Cognitive tasks:

1. Sustained attention and cognitive inhibition The Sustained Attention to Response Task (SART): The SART requires participants to make frequent responses to non-targets and to withhold a response to rarely presented targets. The task simply involves the sequential presentation of 297 single pictures (33 of each kind) presented over 6min. Subjects responded with a key press to each picture, except the 33 occasions when the designated picture appeared (refer to Figure 1). The response required to a non-target stimulus is simply the pressing of a mouse/keyboard, and targets are dispersed randomly in the sequence and occur no more often than 1 in 9 trials on average. In the SART, therefore, commission errors (failure to inhibit responding to a target) or "slips of action" are the result of brief lapses of sustained attention. In the Random SART, the target appears randomly therefore inhibition of a prepotent is essential as the requirement to inhibit a response is unpredictable. Therefore, this task looks at the ability to produce 'correct' inhibitions on inappropriate responses (Robertson et al., 1997).

   The SART has 4 measurable conditions:
   1. Go condition (pressing when required to press)
   2. Omission error (not pressing when required to press)
   3. No-Go condition (not pressing when required to refrain from pressing)
   4. Commission error (pressing when required to refrain from pressing)
2. Working memory The n-back task: The n-back task examines a number of key processes required for working memory. These processes include on-line monitoring, updating information and the manipulation and retention of remembered information. In the task, participants are required to monitor a series of visual stimuli and to indicate when the currently presented stimulus is the same as the one presented n trials (n can be 0, 1, or 2) previously. To begin, in the 0-back condition, participants are required to response to a single pre-determined target picture. In the 1-back condition, the target picture is represented by any picture identical to the immediately preceding one (i.e., one trial back). In the 2-back condition, the target picture is represented by any picture identical to any picture that was presented two trials back. Therefore, the working memory load varies from 0 to 2 items.
3. selective attention and cognitive inhibition The Stroop color and word Task: (Stroop, 1935) The requirements of the Stroop task is to inhibit the more automatic tendency to read a written word while performing the less automatic task of choosing the color of ink in which the word is written, as fast as possible. The participants are required to identify, as quickly as possible, the ink color of the Hebrew words: red, blue, green and yellow, presented in varying colors (red, blue, green and yellow) and press the correct key. The names of the colors will be printed onto keys on the keyboard (i for red, j for yellow, l for blue and m for green). When the participant presses the correct key, reaction time will be recorded, and the next stimulus appeared. Presentation of word stimuli will be divided into blocks, consisting of four blocks of 16 congruent or incongruent (50% each randomly) colored word stimuli. Maximum stimulus duration and interstimulus durations will be 1,300 and 350 msec, respectively. The task procedure is based on previous studies (Peterson et al. 2009).

   Procedural design Parents of children referred to the clinic for ADHD diagnosis and management will be offered to participate in the study. After the parents and participant signed the proper consent form a meeting for evaluation by a psychiatrist will be scheduled. If indeed an ADHD diagnosis is made and methylphenidate treatment is recommended the children will be recruited for the study. The treatment design will be double-blind placebo controlled cross-over. Half of the patients will receive methylphenidate immediate release (IR) first and then placebo and half will receive placebo first and then methylphenidate-IR in a randomized manner. The placebo and methylphenidate-IR pills (identical in appearance) will be placed for each subject in the study group in two cases marked "A" an "B", the content will be written by an RA separately which will decide the order (first placebo or first methylphenidate-IR) using a coin flip, and will be revealed only after the final session and after all questioners will be filled.

   Data analysis

   Data analysis will be made offline:
   * Data preprocessing and artifact correction (using EEGLAB):

   Eye-blink correction Cleaning for movement Filter data • Discrete Regions Analysis (using EEGLAB): Examine the averaged ERP Use t-tests to assess whether the ERP differs across conditions Provide a map of neural response to cognitive tasks • Network analysis (using matlab): Network construction (i.e. nodes, coefficient of cluster, small worldness) Examine network robustness

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents which are being considered for methylphenidate treatment and therefore referred to computerized cognitive tasks with and without methylphenidate IR use as part of their management

Exclusion Criteria:

* study group: Age fewer than 6 and above 18, history of seizure, head trauma, substance abuse or medication other than stimulants, inability to swallow pills.

Exclusion criteria

* control group: Age fewer than 6 and above 18, history of seizure, head trauma, substance abuse, current medication use. Current or lifetime psychiatric disorders.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Complex Network connectivity before treatment - using electrodes signal correlation (P-value) | 0 minutes
  Complex network is measured by metrics that are calculated using graph-theory analysis methods that enable the characterization of the architecture of complex networks. The network is constructed from the EEG signals by correlating the signals between all pairs of electrodes, assuming that each two electrodes that are correlated above a pre-determined threshold are functionally connected and with higher correlation the higher network connectivity. Assessed at baseline before MPH\Placebo according to the above time frames.
Baseline Complex Network connectivity after treatment - using electrodes signal correlation (P-value) | 90 minutes
  Complex network is measured by metrics that are calculated using graph-theory analysis methods that enable the characterization of the architecture of complex networks. The network is constructed from the EEG signals by correlating the signals between all pairs of electrodes, assuming that each two electrodes that are correlated above a pre-determined threshold are functionally connected and with higher correlation the higher network connectivity. Assessed at baseline after MPH\Placebo according to the above time frames.

SECONDARY OUTCOMES:
Complex Network connectivity at Sustained Attention task before treatment - using electrodes signal correlation (P-value) | 11 minutes
  Complex network is measured by metrics that are calculated using graph-theory analysis methods that enable the characterization of the architecture of complex networks. The network is constructed from the EEG signals by correlating the signals between all pairs of electrodes, assuming that each two electrodes that are correlated above a pre-determined threshold are functionally connected and with higher correlation the higher network connectivity. Assessed at Sustained attention task before MPH\Placebo according to the above time frames.
Complex Network connectivity at N-Back task before treatment - using electrodes signal correlation (P-value) | 24 minutes
  Complex network is measured by metrics that are calculated using graph-theory analysis methods that enable the characterization of the architecture of complex networks. The network is constructed from the EEG signals by correlating the signals between all pairs of electrodes, assuming that each two electrodes that are correlated above a pre-determined threshold are functionally connected and with higher correlation the higher network connectivity. Assessed at N-Back task before MPH\Placebo according to the above time frames.
Complex Network connectivity at the Stroop task before treatment - using electrodes signal correlation (P-value) | 30 minutes
  Complex network is measured by metrics that are calculated using graph-theory analysis methods that enable the characterization of the architecture of complex networks. The network is constructed from the EEG signals by correlating the signals between all pairs of electrodes, assuming that each two electrodes that are correlated above a pre-determined threshold are functionally connected and with higher correlation the higher network connectivity. Assessed at the Stroop task before MPH\Placebo according to the above time frames.
Complex Network connectivity at Sustained Attention task after treatment - using electrodes signal correlation (P-value) | 101 minutes
  Complex network is measured by metrics that are calculated using graph-theory analysis methods that enable the characterization of the architecture of complex networks. The network is constructed from the EEG signals by correlating the signals between all pairs of electrodes, assuming that each two electrodes that are correlated above a pre-determined threshold are functionally connected and with higher correlation the higher network connectivity. Assessed at Sustained Attention task after MPH\Placebo according to the above time frames.
Complex Network connectivity at N-Back task after treatment - using electrodes signal correlation (P-value) | 114 minutes
  Complex network is measured by metrics that are calculated using graph-theory analysis methods that enable the characterization of the architecture of complex networks. The network is constructed from the EEG signals by correlating the signals between all pairs of electrodes, assuming that each two electrodes that are correlated above a pre-determined threshold are functionally connected and with higher correlation the higher network connectivity. Assessed at N-Back task after MPH\Placebo according to the above time frames.
Complex Network connectivity at the Stroop task after treatment - using electrodes signal correlation (P-value) | 120 minutes
  Complex network is measured by metrics that are calculated using graph-theory analysis methods that enable the characterization of the architecture of complex networks. The network is constructed from the EEG signals by correlating the signals between all pairs of electrodes, assuming that each two electrodes that are correlated above a pre-determined threshold are functionally connected and with higher correlation the higher network connectivity. Assessed at the Stroop task after MPH\Placebo according to the above time frames.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Gothelf, Prof., Principal Investigator — , . 972-3-5303810
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Rubinson M, Horowitz I, Naim-Feil J, Gothelf D, Moses E, Levit-Binnun N. Electroencephalography Functional Networks Reveal Global Effects of Methylphenidate in Youth with Attention Deficit/Hyperactivity Disorder. Brain Connect. 2019 Jun;9(5):437-450. doi: 10.1089/brain.2018.0630. Epub 2019 May 23. PMID 30919658